CLINICAL TRIAL: NCT05107492
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, THIRD-PARTY OPEN, PLACEBO-CONTROLLED STUDY TO EVALUATE THE PHARMACOKINETICS, SAFETY AND TOLERABILITY FOLLOWING SINGLE SUBCUTANEOUS DOSE OF PF-06480605 IN CHINESE HEALTHY PARTICIPANTS
Brief Title: Evaluation of the Pharmacokinetics, Safety and Tolerability of Single Dose of PF-06480605 in Chinese Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: B7541013
Record Dates: First submitted 2021-11-03; First posted 2021-11-04 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-09

CONDITIONS: Inflammatory Bowel Disease
Keywords: IBD; PK
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): 12 participants will be randomly assigned at an allocation ratio of 3:1 to the active treatment 450mg and placebo arms.
  Interventions: Drug: 450mg; Drug: Placebo
- Cohort 2 (Experimental): 12 participants will be randomly assigned at an allocation ratio of 3:1 to the active treatment 150mg and placebo arms.
  Interventions: Drug: 150mg; Drug: Placebo

INTERVENTIONS:
Drug: 450mg — following a single subcutaneous dose of PF-06480605 450 mg
  Arms: Cohort 1
Drug: 150mg — following a single subcutaneous dose of PF-06480605 150 mg
  Arms: Cohort 2
Drug: Placebo — following a single subcutaneous dose of placebo

SUMMARY:
This is a Phase 1, single-center, randomized, double-blind, third-party open (ie, participant blind, investigator blind and sponsor open), placebo controlled study to investigate PK, safety, tolerability, immunogenicity, and PD of PF 06480605 following a single subcutaneous dose of PF-06480605 450 mg and 150 mg (if needed) in Chinese healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants must be 18 to 45 years of age, inclusive, at the time of signing the ICD.
* Male and female Chinese participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital sign and 12-lead ECG
* BMI of 19 to 27 kg/m2; and a total body weight >50 kg.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* History of HIV infection, hepatitis B, hepatitis C or syphilis; positive testing for HIV, hepatitis B, HCVAb or serological reaction of syphilis.
* History of allergic or anaphylactic reaction to a therapeutic drug.
* History of recent active infections within 28 days prior to the screening visit.
* Participants with a fever within 48 hours prior to dosing.
* History of TB or active or latent or inadequately treated infection.
* Recent exposure to live vaccines within 28 days of the screening visit.
* A positive pregnancy test.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-04-09 (Actual); Study Completion 2022-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7541013

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 12 Chinese healthy adult participants were enrolled, with 9 assigned to PF-06480605 450mg group and 3 to placebo.
Pre-assignment Details: This was a placebo-controlled study of PF-06480605 following 450 mg and 150 mg (if needed) in Chinese healthy adults. Optional 150 mg cohort was not conducted as pharmacokinetic (PK) data of 450mg group did not suggest ethnic difference with previous Western/Japanese studies (by comparing dose-normalized mean exposures/dose-normalized mean concentrations profiles).
Groups:
- PF-06480605 450mg: Participants received a single subcutaneous dose of PF-06480605 450 mg on Day 1.
- Placebo: Participants received matching placebo on Day 1.
Period: Overall Study
Arm/Group | PF-06480605 450mg | Placebo
Started | 9 | 3
Completed (Completion of the entire study including the follow-up phase) | 8 | 3
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received a dose of study intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-06480605 450mg | Placebo | Total
Number analyzed (Participants) | 9 | 3 | 12
Age, Continuous [Median (Full Range); unit: Years] | 34 [23 to 39] | 28 [23 to 40] | 34 [23 to 40]
Age, Customized [Count of Participants; unit: Participants]
  <18 | 0 | 0 | 0
  18-44 | 9 | 3 | 12
  45-64 | 0 | 0 | 0
  >=65 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 8 | 2 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian (Chinese) | 9 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of PF-06480605
Description: Cmax is the maximum observed plasma concentration.
Time Frame: At 0 (prior to dose), 2, 6, 24, 48, 72, 96, 216, 336, 672, 1008, 1344, 2016, and 2712 hours post dose on Day 1
Population: The PK parameter analysis population was defined as all randomized participants who received at least 1 dose of study intervention and for whom at least 1 of the PK parameters of interest was calculated. Data for this outcome measure (OM) was not planned to be collected and analyzed for placebo arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- PF-06480605 450mg: Participants who received PF-06480605 450mg
Arm/Group | PF-06480605 450mg
Number analyzed (Participants) | 9
nanogram per milliliter (ng/mL) | 41530 (26)

2. Primary Outcome: Time for Cmax (Tmax) of PF-06480605
Description: Tmax is the time for Cmax.
Time Frame: At 0 (prior to dose), 2, 6, 24, 48, 72, 96, 216, 336, 672, 1008, 1344, 2016, and 2712 hours post dose on Day 1
Population: The PK parameter analysis population was defined as all randomized participants who received at least 1 dose of study intervention and for whom at least 1 of the PK parameters of interest was calculated. Data for this OM was not planned to be collected and analyzed for placebo arm.
Measure: Median (Full Range); unit: hour
Arm/Group | PF-06480605 450mg
Number analyzed (Participants) | 9
hour | 96.00 [95.9 to 335]

3. Primary Outcome: Area Under the Curve From Time 0 to End of Dosing Interval (AUC14day) of PF-06480605
Description: AUC14day is area under the curve from time 0 to end of dosing interval (Day 14, 336 hours).
Time Frame: At 0 (prior to dose), 2, 6, 24, 48, 72, 96, 216, and 336 hours post dose on Day 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-06480605 450mg
Number analyzed (Participants) | 9
nanogram*hour per milliliter (ng*hr/mL) | 11600000 (26)

4. Primary Outcome: Area Under the Plasma Concentration Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) of PF-06480605
Description: AUCinf is area under the plasma concentration time profile from time 0 extrapolated to infinite time.
Time Frame: At 0 (prior to dose), 2, 6, 24, 48, 72, 96, 216, 336, 672, 1008, 1344, 2016, and 2712 hours post dose on Day 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06480605 450mg
Number analyzed (Participants) | 9
ng*hr/mL | 31390000 (32)

5. Primary Outcome: Terminal Half-life (t1/2) of PF-06480605
Description: t1/2 is the terminal half-life (time required for the plasma concentration to decline by 50%)
Time Frame: At 0 (prior to dose), 2, 6, 24, 48, 72, 96, 216, 336, 672, 1008, 1344, 2016, and 2712 hours post dose on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-06480605 450mg
Number analyzed (Participants) | 9
hour | 306.4 (134.49)

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious AE (SAE) was defined as any untoward medical occurrence that, at any dose: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/incapacity; was a congenital anomaly/birth defect; or other serious situations such as important medical events. TEAEs were events between first dose of study drug and before the end of study (up to follow-up visits). AEs presented below were TEAEs. The investigator was required to use clinical judgment to assess the potential relationship between investigational product and each AE, to define an treatment-related AE.
Time Frame: Day 1 to Day 114
Population: The safety analysis set included all randomized participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants who received placebo
Arm/Group | PF-06480605 450mg | Placebo
Number analyzed (Participants) | 9 | 3
Participants
  All-causality TEAEs | 7 | 3
  Treatment-related TEAEs | 7 | 2

7. Secondary Outcome: Number of Participants With Change From Baseline in Vital Signs Data Meeting the Pre-defined Categorical Summarization Criteria
Description: Vital signs abnormalities included: supine diastolic blood pressure (BP) increase and decrease from BL of >=20mmHg or absolute value <50mmHg; systolic BP increase and decrease from BL of >=30mmHg or absolute value <90mmHg; pulse rate <40 or >120bpm.
Time Frame: From Baseline (BL) to Day 114
Population: The safety analysis set included all randomized participants who received at least 1 dose of study intervention. Participants with evaluable vital signs data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06480605 450mg | Placebo
Number analyzed (Participants) | 9 | 3
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Change From Baseline in Electrocardiogram (ECG) Data Meeting the Pre-defined Categorical Summarization Criteria
Description: ECG assessments included PR, QT, and QTc intervals and QRS complex. ECG abnormalities included PR interval BL >200msec and max >=25% increase from BL, or BL <=200msec and max >=50% increase from BL, or absolute value >=300msec; QRS interval percent change from BL >=50% or absolute value >=140msec, QTcF change from BL >=30msec, or absolute value >450msec.
Time Frame: From BL to Day 114
Population: The safety analysis set included all randomized participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06480605 450mg | Placebo
Number analyzed (Participants) | 9 | 3
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: Safety laboratory assessments included clinical chemistry, hematology, urinalysis, and other tests. Abnormality was determined at the investigator's discretion. Laboratory test abnormalities reported by at least 1 participant are reported in this outcome measure.
Time Frame: From BL to Day 114
Population: The safety analysis set included all randomized participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06480605 450mg | Placebo
Number analyzed (Participants) | 9 | 3
Participants
  Neutrophils > 1.2 x Upper Limit of Normal (ULN) | 1 | 0
  Basophils > 1.2 x ULN | 0 | 1
  Monocytes > 1.2 x ULN | 1 | 0
  Alanine Aminotransferase > 3.0 x ULN | 1 | 0
  Ketones >=1 | 1 | 0

10. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of PF-06480605
Description: AUClast is area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration
Time Frame: At 0 (prior to dose), 2, 6, 24, 48, 72, 96, 216, 336, 672, 1008, 1344, 2016, and 2712 hours post dose on Day 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06480605 450mg
Number analyzed (Participants) | 9
ng*hr/mL | 29990000 (28)

11. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-06480605
Description: Vz/F is the apparent volume of distribution, defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: At 0 (prior to dose), 2, 6, 24, 48, 72, 96, 216, 336, 672, 1008, 1344, 2016, and 2712 hours post dose on Day 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)
Arm/Group | PF-06480605 450mg
Number analyzed (Participants) | 9
liter (L) | 5.839 (42)

12. Secondary Outcome: Apparent Oral Clearance (CL/F) of PF-06480605
Description: CL/F is the apparent oral clearance, which is influenced by the fraction of the dose absorbed. Clearance was estimated from population PK modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: At 0 (prior to dose), 2, 6, 24, 48, 72, 96, 216, 336, 672, 1008, 1344, 2016, and 2712 hours post dose on Day 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/hr)
Arm/Group | PF-06480605 450mg
Number analyzed (Participants) | 9
liter per hour (L/hr) | 0.01434 (32)

13. Secondary Outcome: Number of Participants With Positivie Anti-drug Antibody (ADA) Against PF-06480605
Description: Summary of ADA incidence by visit is presented. ADA positive was defined as titer >=60.
Time Frame: On Days 1 (prior to dose), 15, 29, 57, 85 and 114
Population: The immunogenicity analysis set included all randomized participants who received at least 1 dose of study intervention with at least 1 post-treatment anti-drug (PF-06480605) antibody determination. Number analyzed = Number of participants with observed ADA results at the specific visit.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06480605 450mg
Number analyzed (Participants) | 9
Participants
  Day 1 (Baseline) | 0
  Day 15 | 1
  Day 29 | 4
  Day 57 | 8
  Day 85: number analyzed (Participants) | 6
  Day 85 | 6
  Day 114: number analyzed (Participants) | 7
  Day 114 | 7

14. Secondary Outcome: Number of Participants With Neutralizing Antibody (NAb) Against PF-06480605
Description: Summary of NAb incidence by visit is presented. NAb positive was defined as titer >=5. ADA-positive participants (defined as titer >=60) were analyzed for NAb.
Time Frame: On Days 1 (prior to dose), 15, 29, 57, 85 and 114
Population: The immunogenicity analysis set included all randomized participants who received at least 1 dose of study intervention with at least 1 post-treatment anti-drug (PF-06480605) antibody determination. Number of Participants Analyzed = the total number of participants who had ADA-positive results in this study. Number Analyzed = Number of participants who had ADA-positive results at the specific visit.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06480605 450mg
Number analyzed (Participants) | 9
Participants
  Day 1 (Baseline): number analyzed (Participants) | 0
  Day 1 (Baseline) | 0
  Day 15: number analyzed (Participants) | 1
  Day 15 | 0
  Day 29: number analyzed (Participants) | 4
  Day 29 | 0
  Day 57: number analyzed (Participants) | 8
  Day 57 | 1
  Day 85: number analyzed (Participants) | 6
  Day 85 | 0
  Day 114: number analyzed (Participants) | 7
  Day 114 | 2

15. Secondary Outcome: Total Soluble Tumor Necrosis Factor Like Ligand 1A (sTL1A) Protein Concentration in Serum
Description: The total sTL1A protein concentration in serum is summarized by time.
Time Frame: On Days 1 (prior to dose), 2, 5, 15, 29, 57, 85 and 114
Population: The pharmacodynamic (PD) analysis set included all randomized participants who had at least 1 PD assessment.
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | PF-06480605 450mg | Placebo
Number analyzed (Participants) | 9 | 3
picogram per milliliter (pg/mL)
  Day 1 (Baseline) | 99.7 (15.73) | 89.7 (17.71)
  Day 2 | 314.1 (75.62) | 110.1 (23.46)
  Day 5 | 1470.3 (409.89) | 97.2 (14.39)
  Day 15 | 3817.8 (1172.54) | 116.0 (25.98)
  Day 29 | 3319.2 (2096.47) | 109.6 (13.72)
  Day 57 | 2126.0 (2473.33) | 123.0 (22.61)
  Day 85: number analyzed (Participants) | 6 | 3
  Day 85 | 571.7 (548.71) | 110.9 (22.86)
  Day 114: number analyzed (Participants) | 7 | 3
  Day 114 | 597.6 (404.22) | 108.7 (8.02)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 114
Description: SAEs and nonserious AEs were recorded on the Case Report Form. SAEs were also reported on the Clinical Trial SAE report form to Pfizer Safety within 24h of awareness. The same event may appear as both an AE and SAE. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs/AEs.
Arm/Group | PF-06480605 450mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 7/9 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06480605 450mg (N=9) | Placebo (N=3)
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 1 | 0
Injection site reaction (General disorders) | 5 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 1
White blood cells urine positive (Investigations) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-12-29): https://cdn.clinicaltrials.gov/large-docs/92/NCT05107492/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT05107492/SAP_001.pdf